CLINICAL TRIAL: NCT06909656
Title: Multimodal Electrophysiological Study of Cortico-subcortical Biomarkers of Tics in Tourette Syndrome
Acronym: BioTic
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2023/84
Record Dates: First submitted 2025-03-24; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Tourette Syndrome
Keywords: Tourette Syndrome; Local field potentials; Deep Brain Stimulation
MeSH Terms: conditions — Tourette Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with Tourette's syndrome (Experimental): Patient with Tourette's syndrome receiving deep brain stimulation treatment with implantation of the PERCEPT™ device as part of their medical management.
  Interventions: Other: Multimodal electrophysiological recordings

INTERVENTIONS:
Other: Multimodal electrophysiological recordings — Intervention(s): Multimodal electrophysiological recordings (Local field potentials, High-Resolution Electroencephalogram, Electromyogram) coupled with video analysis, in experimental condition, in uncontrolled tic and voluntary ("tic-like") movement.

SUMMARY:
Tourette syndrome (TS) is a complex neurodevelopmental disorder characterized by the occurrence of involuntary movements (motor tics) and vocalizations (phonic tics). The onset of TS is usually in childhood, and the prevalence of TS is estimated between 0.3 and 0.9% before the age of 18, decreasing progressively after that age. Most patients also suffer from associated psychiatric comorbidities (ADHD, OCD, mood disorders). Although the cause of TS remains unknown, the preferred hypothesis is the interaction of predisposing genetic factors and precipitating environmental factors (perinatal accidents, infectious diseases). From a pathophysiological point of view, it is widely demonstrated by structural, electrophysiological studies, functional neuroimaging, as well as by different animal models, that dysfunctions of the cortico-striato-pallido-thalamo-cortical loops (responsible for the regulation of movements, cognitive processes, and emotions) play a major role in the genesis of tics. Deep brain stimulation (DBS) treatment can be proposed as an invasive therapy in patients with severe TS resistant to usual treatments (psychotherapy, pharmacological treatments). In a well-selected population of drug-resistant patients, DBS allows an estimated overall improvement of 30 to 50% in the YGTSS score. The deep brain stimulation method currently used in TS is based on continuous (24/7) and undifferentiated stimulation (fixed electrical intensity). This stimulation paradigm, devoid of adaptability to the patient's symptoms, could be at the origin of undesirable effects (related to the modulation of physiological signals), of a sub-optimal efficiency, or of an unnecessary overuse of the stimulator's capacities (battery depletion). The development of new deep brain stimulation paradigms ("closed-loop stimulation"), allowing the identification of pathological neuronal activity and the dynamic adaptation of stimulation parameters to these neuronal signals, requires reliable and reproducible pathological biomarker, correlated with the occurrence of tics.

However, in TS, electrophysiological abnormalities are still not well characterized, and most of the work published on the subject were based on intraoperative recordings and needs to be confirmed on recordings at a distance from the surgery before its potential use in closed-loop stimulation paradigms. Indeed, during the first weeks after surgery, different factors tend to modify the electrophysiological signals.

Several questions arise at the end of this healing period:

* Are these pathological oscillations (distinct from the brain oscillations induced by physiological voluntary movement) still detectable weeks after the surgery?
* What are the temporal dynamics of these oscillations around a tic?
* What is the spatial topography of these oscillations within the GPi?
* Is there a strong inter-individual variability?
* How are changes in cortical activity associated with these subcortical oscillations?
* Are the modulations of pallidal activity alone sufficient to predict the occurrence of a tic? Thus, our study aims to define precisely the cortico-subcortical activity concomitant with the occurrence of a tic, and to identify reliable and reproducible biomarker(s) associated with tics in TS.

In order to specify these biomarker(s), their temporal correlation to tic occurrence, their spatial distribution, as well as the dynamics and cortico-subcortical coherence of the identified abnormalities, we propose a prospective study on 10 patients with severe and drug-resistant TS, treated by bi-pallidal deep brain stimulation as part of routine care (no device implantation as part of the research).

An evaluation of pallidal LFP synchronized with a high-resolution video-electroencephalography recording (128 to 256 sensors) will be performed at a distance (M+[3-48]) from surgery, in order to determine the variations in pallidal and electroencephalographic activity surrounding the occurrence of tics. A control condition with voluntary ("tic-like") movement will be carried out in a second time, to distinguish the modifications related to the voluntary movement from those related to the occurrence of a tic. A reconstruction of the electrode positioning will be performed using the LeadDBS pipeline, and individual and group analyses will be performed to specify the mapping of pathological oscillations within the pallidum and throughout the cerebral cortex.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 16 years old.
* Disabling and drug-resistant Tourette's syndrome.
* Receiving deep brain stimulation treatment with implantation of the PERCEPT™ Device as part of their medical management.
* Normal brain MRI.
* Subject affiliated or beneficiary of a social security system.
* Free and informed consent of the patient and, for minors, of the minor and at least one parental authority.

Exclusion Criteria:

* Major depressive syndrome (Beck Depression Inventory (BDI-II) > 20).
* MRI showing significant brain atrophy or significant hyperintensities.
* Pregnant or nursing mothers.
* Person unable to give personal consent.
* Person subject to a legal protection measure (curatorship, guardianship) or placed under court protection.
* Patient included in another research protocol with an interdiction of participation to another research or in an exclusion period

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-02-17 (Estimated); Study Completion 2027-02-17 (Estimated)

PRIMARY OUTCOMES:
Spectral power | Inclusion visit
  Pallidal spectral power in the 2 clinical conditions (i) Tic [pre-tic-post] and (ii) Voluntary ("tic-like") movement [pre-movement-post] respectively.

SECONDARY OUTCOMES:
Electrode localization | Inclusion visit
Pallidal and cortical spectral power | Inclusion visit
  Pallidal and cortical spectral power analysis in the 2 clinical conditions (i) Tic and (ii) Voluntary movement ("tic-like").
Pallidal and cortical time-frequency | Inclusion visit
  the 2 clinical conditions (i) Tic and (ii) Voluntary movement ("tic-like").
Cortico-subcortical coherence | Inclusion visit
  Cortico-subcortical coherence of the recorded oscillations.
Cortico-subcortical phase synchronization | Inclusion visit
  Cortico-subcortical phase synchronization of the recorded oscillations.
Cortico-subcortical phase-amplitude coupling | Inclusion visit
  Cortico-subcortical phase-amplitude coupling of the recorded oscillations.
Adult ADHD Self-Report Scale (ASRS) Score | Inclusion visit
  Used to assess symptoms of Attention-Deficit/Hyperactivity Disorder (ADHD) in adults, it consists of 18 items.
  Total score of 0 to 14: Low probability of ADHD.
  Total score of 15 to 24: Intermediate probability that the person exhibits symptoms of ADHD.
  Total score of 25 to 36: Suggests a high probability of ADHD.
Adult ADHD Self-Report Scale (ASRS) Score | One month before inclusion
  Used to assess symptoms of Attention-Deficit/Hyperactivity Disorder (ADHD) in adults, it consists of 18 items.
  Total score of 0 to 14: Low probability of ADHD.
  Total score of 15 to 24: Intermediate probability that the person exhibits symptoms of ADHD.
  Total score of 25 to 36: Suggests a high probability of ADHD.
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) Score | Inclusion visit
  Considered as the reference scale for evaluating obsessive-compulsive disorders. Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is designed to assess both the types of symptoms and their severity. The Y-BOCS evaluates 10 items, each rated from 0 (no symptoms) to 4 (extreme symptoms).
  The total score ranges as follows:
  0 to 7: Normal
  8 to 15: Mild
  16 to 23: Moderate
  24 to 31: Severe
  32 to 40: Very severe
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) Score | One month before inclusion
  Considered as the reference scale for evaluating obsessive-compulsive disorders. Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is designed to assess both the types of symptoms and their severity. The Y-BOCS evaluates 10 items, each rated from 0 (no symptoms) to 4 (extreme symptoms).
  The total score ranges as follows:
  0 to 7: Normal
  8 to 15: Mild
  16 to 23: Moderate
  24 to 31: Severe
  32 to 40: Very severe
Yale Global Tic Severity Scale (YGTSS) Score | Inclusion visit
  semi-structured clinical interview scale that is considered the gold standard for assessing the severity of tics in both children and adults. The YGTSS evaluates the number, frequency, intensity, complexity, and distress associated with motor and vocal tics over the past week. Each domain is assessed on a 6-point scale (from 0 to 5), with a separate, more global score for "overall disability" concerning the individual's daily life and activities.
  Five sub-scores can be extracted:
  The total "motor tic" score (from 0 to 25)
  The total "vocal tic" score (from 0 to 25)
  The total "tic" score (sum of the two previous scores)
  The overall disability assessment (one item; from 0 to 50)
  The global severity score (from 0 to 100)
Yale Global Tic Severity Scale (YGTSS) Score | One month before inclusion
  semi-structured clinical interview scale that is considered the gold standard for assessing the severity of tics in both children and adults. The YGTSS evaluates the number, frequency, intensity, complexity, and distress associated with motor and vocal tics over the past week. Each domain is assessed on a 6-point scale (from 0 to 5), with a separate, more global score for "overall disability" concerning the individual's daily life and activities.
  Five sub-scores can be extracted:
  The total "motor tic" score (from 0 to 25)
  The total "vocal tic" score (from 0 to 25)
  The total "tic" score (sum of the two previous scores)
  The overall disability assessment (one item; from 0 to 50)
  The global severity score (from 0 to 100)

CONTACTS AND LOCATIONS:
Overall Officials: Edouard COURTIN, Dr, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No